CLINICAL TRIAL: NCT05710276
Title: Assessment of Intestinal Inflammation by Infrared Thermography in Pediatric Crohn Disease
Acronym: THERMO-CROHN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: PI2022_843_0001
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Crohn Disease; Infrared Thermography; Child
Keywords: Crohn Disease; Infrared thermography; Faecal Calprotectin; PCDAI; Child
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: abdominal infrared radiation — In a specific room (controlled temperature and humidity) with a patient lying on his back, we will determine the abdominal infrared radiation with a FLIR® thermal camera (without contact) and quantify the thermal signal by spectral analysis (in degrees Celsius).

SUMMARY:
The assessment of digestive inflammation and disease activity in paediatrics Crohn's disease (CD) is currently based on anamnestic, clinical and paraclinical elements such as the paediatric CD activity index (wPCDAI) , faecal calprotectin measuring or digestive endoscopy. Infrared thermal imaging is based on capturing electromagnetic waves, on a specific Wavelength, emitted by the human body surface and representing local thermic-metabolic activity. It concern metabolic activity in digestive inflammations. Infrared imaging is a non-invasive, contactless, stressless technique that assess the variations in skin surface temperature of the patient's entire abdomen or more targeted areas in a single photography. This technique would be useful for determination of Crohn's disease activity, inflammation's degree and partial mapping of inflammatory lesions.

In a specific room with a patient lying, the investigators will determine the abdominal infrared radiation with a FLIR® thermal camera. This will be correlated with the measurement of the faecal calprotectin concentration and the composite CD activity index wPCDAI.

All measurements will be performed during the standard follow-up of Crohn disease. No additional follow will be necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CD according to the Porto criteria [6]
* Aged from 4 years to 17 years-old
* Follow-up at the Amiens Picardie University Hospital (CHU Amiens Picardie)
* Child's affirmative agreement and assent and permission of their parents to participate in research

Exclusion Criteria:

* Recent abdominal surgery
* Other Inflammatory bowel disease

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
correlation between the quantification of abdominal infrared radiation and faecal calprotectin concentration | one year
  correlation between the quantification of abdominal infrared radiation determined by the FLIR® thermal camera and quantified by the spectral analysis of the thermal signal (in degrees Celsius) and the determination of faecal calprotectin concentration (µg/g of faeces). This concentration will be determined by ELISA method at Biochemistry in Amiens Picardie Faculty hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No